CLINICAL TRIAL: NCT00811902
Title: A 14-Week, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy, Safety, and Tolerability of Nerispirdine 50 mg, 100 mg, and 200 mg in Patients With Multiple Sclerosis.
Brief Title: Efficacy, Safety, and Tolerability of Nerispirdine in Patients With Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DRI10566; 2008-001999-67 (EudraCT Number)
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — nerispirdine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Nerispirdine 50mg (Experimental): Nerispirdine 50mg once daily for 14 weeks
  Interventions: Drug: Nerispirdine
- Nerispirdine 100mg (Experimental): Nerispirdine 100mg once daily for 14 weeks
  Interventions: Drug: Nerispirdine
- Nerispirdine 200mg (Experimental): Nerispirdine 200mg once daily for 14 weeks
  Interventions: Drug: Nerispirdine
- Placebo (Placebo Comparator): Placebo for Nerispirdine once daily for 14 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Nerispirdine — tablet, oral administration
  Other Names: HP184
  Arms: Nerispirdine 100mg; Nerispirdine 200mg; Nerispirdine 50mg
Drug: placebo — tablet, oral administration
  Arms: Placebo

SUMMARY:
The primary objective is to assess the activity of nerispirdine in improving the ability to walk, in patients with multiple sclerosis (MS).

Secondary objectives:

* To assess other measures of walking ability, tiredness, and lower limb muscular strength, spasticity, clinical assessment by subject and clinical assessment of change by the Study Investigator
* To assess the safety and tolerance of nerispirdine
* To evaluate the pharmacokinetics (PK) parameters of nerispirdine

DETAILED DESCRIPTION:
Total duration per patient is approximately 19 weeks in total, comprising a 3-week screening period inclusive of a 2-week placebo run-in period, a 14-week treatment period, and a 2-week placebo run-out (follow-up) period

ELIGIBILITY:
Inclusion Criteria:

* Clinically definite MS (according to McDonald criteria),

Exclusion Criteria:

* Multiple sclerosis exacerbation or clinical relapse within 6-month prior to the screening visit.
* Subject who is not able to complete two trials of a timed 25 foot walk, with or without an assisted device,
* Patients without valid V1, V2, and V4 T25-FW measurements are not eligible for randomization.
* Female patients who are either pregnant or breastfeeding.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2008-12; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Responder criterion based on consistency of improved response in walking speed on the Timed 25-Foot Walk (T25-FWT) | 14 weeks

SECONDARY OUTCOMES:
Change from baseline to endpoint in the 12-item MS Walking Scale (MSWS-12) | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (7):
- Sanofi-aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-aventis Administrative Office, Laval, Canada
- Sanofi-aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Lysaker, Norway
- Sanofi-aventis Administrative Office, Barcelona, Spain